CLINICAL TRIAL: NCT06943092
Title: Efficacy of Piroxicam Versus Diclofenac as Components of Multimodal Analgesic for Post Caesarean Section Analgesia.
Brief Title: Piroxicam Versus Diclofenac for Post Caesarean Section Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Teaching Hospital Abakaliki (Other Government)
Responsible Party: Principal Investigator, Assumpta Nnenna Nweke, Principal Investigator, Federal Teaching Hospital Abakaliki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FETHA/REC/VOL2/2019/293
Record Dates: First submitted 2025-04-14; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Analgesia; Post Caserean
Keywords: Pentazocine; Piroxicam; Diclofenac; Post caesarean analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Open label randomised controlled trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piroxicam group (Experimental): Group A received a single dose of intramuscular Piroxicam 20 mg.The first dose was administered immediately after skin closure. Thereafter, this group received intramuscular Pentazocine 30mg 6 hourly for 24 hours.
  Interventions: Drug: Piroxicam group
- Diclofenac group (Active Comparator): Group B received two doses of intramuscular diclofenac 75 mg.The first dose was administered immediately after skin closure and the second dose was administered 12 hours after the first dose. intramuscular Pentazocine 30mg was given 6 hourly for 24 hours.
  Interventions: Drug: Diclofenac group

INTERVENTIONS:
Drug: Piroxicam group — Experimental drug
  Arms: Piroxicam group
Drug: Diclofenac group — Active drug
  Arms: Diclofenac group

SUMMARY:
Multimodal analgesic combination of pentazocine-diclofenac has been found to be superior to pentazocine-piroxicam and was associated with a higher level of maternal satisfaction. our study aims to determine the efficacy of piroxicam when compared with diclofenac as pain relief post caesarean section.

DETAILED DESCRIPTION:
ABSTRACT Background: Postoperative pain is unavoidable after caesarean section. It constitutes a big challenge to patient's recovery and maternal-infant bonding. The importance of adequate pain control cannot be over emphasized but there is no gold standard for post caesarean section analgesia. A multimodal approach to post caesarean section pain control has been shown to enhance analgesia and reduce side effects but the right combination of analgesics is yet to be determined.

Objective: To compare the efficacy of Pentazocine and Piroxicam versus Pentazocine and Diclofenac for post caesarean section analgesia within first 24 hours.

Method: Eligible participants undergoingelective caesarean section atAlex Ekwueme Federal University Teaching Hospital Abakaliki (AEFUTHA) and St Patrick's Mile 4 Hospital Abakaliki were randomized into two groups, A and B, of 54 participants each using computer generated list of random numbers. Group A receiveda single dose of intramuscular Piroxicam 20mg, while group B received two doses of intramuscular Diclofenac 75mg given 12 hours apart. Participants in both groups also received intramuscular Pentazocine 30mg 6 hourly for 24 hours. The first dose of the drugs was administered immediately after skin closure. The primary outcome measure was control of postoperative painwithin the first 24 hours after caesarean section assessed using visual analogue scale, while the secondary outcome measures were the maternal drug side effects (epigastric pain, nausea etc) and participants' satisfaction. Data obtained was entered into a predesigned sheet and analyzed using Statistical Package for Social Science (IBM SPSS) software (version 24, Chicago II, USA). A difference with a p-value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women carrying live singleton fetusesat 37-42 weeks' gestational age.
* Consentingparturients who had elective caesarean section, under spinal anaesthesia.
* American Society of Anaesthesiologists (ASA) I-II physical status.

Exclusion criteria

* Caesarean sections under general or epidural anesthesia
* Known allergy to Pentazocine, Diclofenacand or Piroxicam
* Patients with uncontrolled hypertension/ pre-eclampsia or eclampsia
* Multiple gestation
* History of peptic ulcer disease,asthma
* Patients with chronic pain or on long term opioids
* Women with dead fetuses or fetuses with congenital abnormalities
* Patients who are unable to rate the pain due to psychiatric illness or illiteracy.
* Parturients with severe obstetric haemorrhage, and sickle cell haemoglobinopathy
* Those that declined consent to participate in the study despite adequate counselling.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 108 (Actual)
Dates: Start 2020-01-11 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours
  This is the post operative pain within the first 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Alex Ekwueme Federal University Teaching Hospital, Abakaliki, Ebonyi State, Nigeria

IPD SHARING:
Plan to Share IPD: No
This will be following publication